CLINICAL TRIAL: NCT06961942
Title: Enhancing Endoscopic Scoring Consistency and Accuracy in IBD: a Video-based Training Approach
Acronym: CONCORDIA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CONCORDIA
Record Dates: First submitted 2025-04-07; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: IBD (Inflammatory Bowel Disease)
Keywords: Training; Scoring; IBD
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: The CONCORDIA study will be conducted in three sequential time periods. During Time Period 1 (two months), all participants will independently score 15 endoscopic videos using the updated Rutgeerts score and 15 videos with ePDAI and SES-pouch, supplemented with a general Visual Analogue Scale (VAS) score (0=no inflammation, 10=most severe inflammation). No specific guidance will be provided during that phase.
  Following the first video assessment only participants in Group A will attend the structured training module.
  During Time Period 2 (one month), all participants will score the same 15 + 15 videos. However, only participant in Group A will have access to the explanatory videos used in the online training module.
  After the second video assessment participants in Group B will receive the structured training module.
  During Time Period 3 (one months), participants in Group B will score the 15 + 15 videos again while having access to the explanatory videos used in the online training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Early training) (Active Comparator): Following the first video assessment only participants in Group A will attend the structured training module.
  During Time Period 2 (approximately one month), all participants will score the same 15 + 15 videos. However, only participant in Group A will have access to the explanatory videos used in the online training module.
  Interventions: Other: Training
- Group B (Late training) (No Intervention): After the second video assessment participants in Group B will receive the structured training module.
  During Time Period 3 (approximately one month), participants in Group B will score the 15 + 15 videos again while having access to the explanatory videos used in the online training module.

INTERVENTIONS:
Other: Training — A structured teaching module for fellows in training will be prepared and conducted at three university centres, namely University Hospitals Leuven, Ljubljana University Medical Centre, and CHU de Bordeaux. The training module will include short endoscopic videos (different from the pre- and post-training set), which participants will score in real-time using a polling application. This will be followed by a step-by-step demonstration of each scoring principle with explanations of the reasoning behind specific scores. Each scoring system will be reviewed in a short training video that provides a structured demonstration, highlights common pitfalls, and showcases typical IBD-associated endoscopic features. After the video training, participants will have the opportunity to ask questions to the experts.
  Arms: Group A (Early training)

SUMMARY:
Endoscopic scoring systems are vital for the objective assessment of disease activity being used in both clinical trials and daily clinical practice. These standardized scoring systems are essential for diagnosing, evaluating endoscopic healing, monitoring treatment response, and predicting clinical outcomes.

One of the primary challenges in implementing these scoring systems is inter-observer variability, as highlighted by significant discrepancies between scores assigned by local and central reviewers. However, the performance of these systems among experts has been shown to be excellent, suggesting that achieving consistent and accurate scoring requires a high level of exposure and proficiency.

Inconsistent scoring, especially among less experienced clinicians, poses a challenge to the reliability of these scoring systems.

The primary objective of this study is to evaluate the improvement of scoring accuracy after training with structured educational videos with a specific focus on the learning curve and the practical application of endoscopic scoring systems.

DETAILED DESCRIPTION:
Endoscopy is a cornerstone in diagnosis, management and monitoring of patients with inflammatory bowel disease (IBD), comprising Crohn's disease (CD) and ulcerative colitis (UC). Endoscopy in combination with histological assessment plays a crucial role in diagnosis of IBD, distinguishing between UC and CD and ruling out other diseases with similar clinical presentations. The STRIDE-II consensus, developed by the International Organization for the Study of IBD (IOIBD), highlights endoscopic healing as the primary long-term therapeutic goal. Achieving endoscopic healing is associated with improved patient outcomes, including steroid-free remission, a reduced risk of clinical relapse, hospitalization, colectomy, and dysplasia or colorectal cancer.

Endoscopic scoring systems are vital for the objective assessment of disease activity being used in both clinical trials and daily clinical practice. These standardized scoring systems are essential for diagnosing, evaluating endoscopic healing, monitoring treatment response, and predicting clinical outcomes.

The most widely adapted scoring systems in IBD include:

* The Simple Endoscopic Score for Crohn's Disease (SES-CD) evaluates four key parameters: ulcer size, ulcerated surface, affected surface area, and luminal narrowing. It offers a straightforward, clinically validated scoring system that strongly correlates with indices such as the Crohn's Disease Activity Index.
* The updated Rutgeerts Score provides accurate and clinically relevant assessments of postoperative recurrence in CD and facilitates the prediction of clinical and surgical outcomes for patients with an ileocolonic anastomosis.
* The Endoscopic Mayo Score is a component of the broader Mayo scoring system used to assess disease activity in UC. It evaluates the extent and severity of mucosal inflammation, correlating well with clinical outcomes, including treatment response.
* The Ulcerative Colitis Endoscopic Index of Severity (UCEIS) standardizes the evaluation of endoscopic severity in UC. It incorporates more detailed descriptors of mucosal appearance, including vascular pattern, bleeding, erosions, and ulcerations to describe overall disease severity (Neurath & Travis, 2012).
* The Pouchitis Disease Activity Index (PDAI) assesses pouchitis severity using clinical symptoms, endoscopic findings, and histological features of the pouch. This quantitative tool helps to diagnose and monitor pouchitis. Endoscopic part of PDAI (ePDAI) consists of six features describing mucosal changes: oedema, granularity, friability, loss of vascular pattern, mucous exudate and ulceration.
* The Simplified Endoscopic Score for Pouchitis (SES-pouchitis), recently suggested as an alternative to the PDAI, adapts the SES-CD framework to focus on one single segment, namely the ileal pouch.

One of the primary challenges in implementing these scoring systems is inter-observer variability, as highlighted by significant discrepancies between scores assigned by local and central reviewers. However, the performance of these systems among experts has been shown to be excellent, suggesting that achieving consistent and accurate scoring requires a high level of exposure and proficiency.

Inconsistent scoring, especially among less experienced clinicians, poses a challenge to the reliability of these scoring systems. Daperno et al. demonstrated in their study that a structured educational training program significantly enhanced inter-observer agreement. The study, including 237 gastroenterologists with at least three years of post-certification experience, showed substantial improvements in scoring consistency across multiple IBD scoring systems (SES-CD, Mayo Endoscopic Subscore, and Rutgeerts Score) following the training. These findings emphasize the importance of comprehensive training to ensure reliable and consistent endoscopic evaluations. Intensive education programs are crucial for improving scoring accuracy, enabling effective disease monitoring and management in IBD.

New scoring systems for assessing disease activity are developing, however, they are relatively unknown among gastroenterologists and are not yet widely used in clinical practice.

In the CONCORDIA study, the investigators will evaluate gastroenterology fellows' familiarity with these new scoring systems and assess whether structured endoscopic video assisted training improves scoring accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Gastroenterology fellows

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Improvement of Updated Rutgeerts scoring accuracy after training with structured educational videos | 3 months
  In substudy A, the investigators will focus on the updated Rutgeerts score for patients with Crohn's disease that previously underwent an ileocolonic resection with ileocolonic anastomosis.
Improvement of ePDAI scoring accuracy after training with structured educational videos | 3 months
  In substudy B, the investigators will focus on the Endoscopic element of the Pouchitis Disease Activity Index (ePDAI) for patients with ulcerative colitis that previously underwent a proctocolectomy with ileal pouch-anal anastomosis (IPAA).
  ePDAI consists of six features describing mucosal changes: oedema, granularity, friability, loss of vascular pattern, mucous exudate and ulceration.
IImprovement of SES-pouchitis scoring accuracy after training with structured educational videos | 3 months
  In substudy B, the investigators will focus on the Simple Endoscopic Score (SES)-pouchitis for patients with ulcerative colitis that previously underwent a proctocolectomy with ileal pouch-anal anastomosis (IPAA).
  SES-pouchitis evaluates four key parameters, ulcer size, ulcerated surface, affected surface area, and luminal narrowing, in the ileal pouch.

IPD SHARING:
Plan to Share IPD: No
The primary objective of this study is to set-up a training for gastroenterology fellows